CLINICAL TRIAL: NCT02050880
Title: Crossed Precision Design Study of the Nidek Optical Coherence Tomography RS-3000, RS-3000 Lite and RS-3000 Advance for the Measurements of Retinal and RNFL Thickness, Optic Disc Analysis, and Pachymetry
Brief Title: OCT Agreement and Crossed Precision Study
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: RS-3000 series Protocol 1
Record Dates: First submitted 2014-01-22; First posted 2014-01-31 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Glaucoma; Retinal Disease; Corneal Disease
Keywords: Normal Eyes; Eye; Disorder with Glaucoma; Eye; Disorder with Retinal Disease; Eye; Disorder Corneal Disease incl kerato-refractive group
MeSH Terms: conditions — Glaucoma; Retinal Diseases; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal eyes: Eyes without pathology.
- Glaucoma: Eyes with Glaucoma.
- Retinal: Eyes with Retinal Disease.
- Corneal: Eyes with corneal disease including a kerato-refractive group.

SUMMARY:
The purpose of this study is to asses the agreement of the RS-3000 Lite and RS-3000 Advance to the RS-3000, assess the crossed precision of each study device and to assess the transference of a reference database from the RS-3000 to the RS-3000 Lite and to the RS-3000 Advance.

ELIGIBILITY:
Inclusion Criteria: NORMAL EYES

* Subjects who do not have pathology in both eyes

Inclusion Criteria: GLAUCOMA

* Subjects who have a glaucoma diagnosis

Inclusion Criteria: RETINAL

* Subjects who have a retinal diagnosis including but not limited to:

  1. Diabetic macular edema
  2. Dry age related macular degeneration
  3. Wet age related macular degeneration
  4. Cystoid macular edema
  5. Epiretinal membrane
  6. Macular hole

Inclusion Criteria: CORNEAL

* Subjects who has one of these diagnosis:

  1. Post status LASIK surgery
  2. Keratoconus
  3. Other corneal dystrophies or degenerations.

Exclusion Criteria: ALL EYES

* Subjects who have any of the following conditions

  1. Diabetes mellitus (DM) and/or diabetic retinopathy
  2. Uncontrolled Hypertension (HT)
  3. Cerebral infarction, cerebral hemorrhage, cranial nerve neoplasm and other central nervous system diseases affecting vision
  4. Cardiac, hepatic, renal and hematologic diseases
  5. A current condition requiring systemic administration of steroid
  6. A history of, or currently receiving, anticancer therapy
  7. Epileptic seizures which are optically induced
  8. Dementia
* Subjects who have other life threatening and debilitating systemic diseases

Note: Additional criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinic subjects, general population
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | Approximately four hours
  Time frame is the maximum duration of hospital stay
Optic Disc Analysis | Approximately four hours
  Time frame is the maximum duration of hospital stay
Corneal Thickness | Approximately four hours
  Time frame is the maximum duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global Opthalmology Research Center, Santa Ana, California, United States